CLINICAL TRIAL: NCT02112799
Title: A Phase 1 Dose-Ranging Study to Assess the Safety, Pharmacokinetics and Initial Antiviral Efficacy of NVR 3-778 in Healthy Volunteers and Patients With Chronic Hepatitis B
Brief Title: Safety and Efficacy Study of NVR 3-778 in Healthy Volunteers and Hepatitis B Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novira Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: NVR3-778-101
Record Dates: First submitted 2014-04-09; First posted 2014-04-14 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — NVR 3-778; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NVR 3-778 (Experimental): NVR 3-778 in varying doses of capsules by mouth for 1 day, 14 days, or 28 days
  Interventions: Drug: NVR 3-778
- Placebo for NVR 3-778 (Placebo Comparator): Placebo for NVR 3-778 in varying doses of capsules by mouth for 1 day, 14 days, or 28 days
  Interventions: Drug: Placebo for NVR 3-778
- NVR 3-778 and Pegasys (Experimental): NVR 3-778 and Pegasys in combination in a yet to be determined dose by mouth and subcutaneous injection for 28 days
  Interventions: Drug: NVR 3-778; Drug: Pegasys
- Pegasys (Active Comparator): Pegasys alone in a yet to be determined dose by subcutaneous injection for 28 days
  Interventions: Drug: Pegasys

INTERVENTIONS:
Drug: NVR 3-778
  Arms: NVR 3-778; NVR 3-778 and Pegasys
Drug: Placebo for NVR 3-778 — Sugar pill manufactured to mimic the NVR 3-778 capsule
  Arms: Placebo for NVR 3-778
Drug: Pegasys
  Other Names: peginterferon alfa-2a
  Arms: NVR 3-778 and Pegasys; Pegasys

SUMMARY:
This Phase 1 trial will assess the dose-related safety and PK profile of different doses of NVR 3-778, first in healthy volunteer subjects (part I) and subsequently in patients with chronic hepatitis B (part II). Additionally, in Part II, changes in patients' serum HBV DNA levels and other virologic efficacy parameters will be assessed.

DETAILED DESCRIPTION:
The Part I (Phase 1a) assessments of the dose-related safety and PK of NVR 3-778 in volunteers will be conducted an established Phase 1 unit, which will facilitate the overnight confinements and frequent safety assessments and blood sampling required for the Part I evaluations. The Part II (Phase 1b) assessments of the dose-related safety, PK, and initial antiviral efficacy of NVR 3-778 in hepatitis B patients will also be conducted at approximately 14 different sites to meet enrollment goals of 54-84 chronic hepatitis B patients.

To promote objective safety and tolerance assessments during this trial, study subjects, and site personnel administering the study drug and performing the clinical assessments on the subjects, will be blinded to individual subjects' treatments assignments (active NVR 3-778 or placebo doses), for all treatment cohorts in the study. Study advancement to subsequent volunteer cohorts in Part I and subsequent patient cohorts in Part II will require satisfactory interim reviews of available cumulative safety data by the Part I and Part II Safety Review Committees (SRCs), using the safety criteria and review procedures described in the protocol. Also, there will be two interim reviews of safety data by an independent Safety Monitoring Board (SMB), as described in the protocol.

ELIGIBILITY:
Healthy volunteers may be male or female between 18 and 65 years old with a BMI of 18-32kg/m2. They must be in good health not have any health condition which could interfere with the absorption, distribution or elimination of study drug, or with the clinical and laboratory assessments in this study.

Patients enrolling in Part II of the study, may be male or female between 18 and 65 years of age, with a BMI of 18-35kg/m2. Patients must have HBeAg positive, chronic hepatitis B with no history of clinical decompensation, and must not have been treated for hepatitis B before.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-04-30 (Actual); Primary Completion 2016-05-18 (Actual); Study Completion 2016-05-18 (Actual)

PRIMARY OUTCOMES:
To assess the dose-related safety and tolerability of NVR 3-778 in healthy volunteers and hepatitis B patients | Up to 28 days

CONTACTS AND LOCATIONS:
Locations (2):
- New Zealand (2):
  - Hamilton, Waikato Region
  - Auckland

REFERENCES:
- [Derived] Yuen MF, Gane EJ, Kim DJ, Weilert F, Yuen Chan HL, Lalezari J, Hwang SG, Nguyen T, Flores O, Hartman G, Liaw S, Lenz O, Kakuda TN, Talloen W, Schwabe C, Klumpp K, Brown N. Antiviral Activity, Safety, and Pharmacokinetics of Capsid Assembly Modulator NVR 3-778 in Patients with Chronic HBV Infection. Gastroenterology. 2019 Apr;156(5):1392-1403.e7. doi: 10.1053/j.gastro.2018.12.023. Epub 2019 Jan 6. PMID 30625297